CLINICAL TRIAL: NCT01781806
Title: A Pilot Demonstration Project to Operationalize Pre-exposure Prophylaxis as Part of Combination HIV Prevention Among Men Who Have Sex With Men (MSM) and Transgender Women in Los Angeles County
Brief Title: A Demonstration Project to Add Pre- or Post-exposure Prophylaxis to Combination HIV Prevention Services
Acronym: PATH-PrEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government); Los Angeles LGBT Center (Other); The OASIS Clinic (Unknown); AIDS Project Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Raphael Landovitz, Principal Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EI11-LA-002
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort H (PrEP) (Active Comparator): Participants in the H cohort will be provided with a CPP, including daily oral emtricitabine/tenofovir-based PrEP.
  High Risk Cohort Criteria (one or more of the following has to be met):
  1. No condom use during anal intercourse with ≥3 male sex partners who are HIV-positive or of unknown HIV status during the last three months.
  2. STD diagnosis during the last 12 months.
  3. Previous PEP use during the last 12 months (* see exclusion criteria)
  4. Has at least one HIV infected sexual partner for ≥4 weeks.
  Interventions: Drug: emtricitabine 200mg/tenofovir 300mg
- Cohort LM (PEP) (Active Comparator): Participants who do not meet criteria for High Risk (Cohort H) will be assigned to the LM (low moderate) cohort and will receive a customized prevention package based on baseline assessments (in the same manner as the Cohort H Participants). In addition, they will receive education on the availability and use of post-exposure prophylaxis.
  Interventions: Drug: emtricitabine 200mg/tenofovir 300mg

INTERVENTIONS:
Drug: emtricitabine 200mg/tenofovir 300mg — The intervention medication will be tenofovir + emtricitabine, provided as a fixed-dose combination tablet as Truvada®. Dosing is 1 tablet by mouth once daily. For participants with a a confirmed (i.e. two consecutive) reduction in creatinine clearance (CrCl) to <50 mL/min, Truvada will be dose-reduced to 1 tablet by mouth every other day. For patients with CrCl <30 mL/min, Truvada will be discontinued.
  Other Names: Truvada

SUMMARY:
The purpose of this study is to evaluate the safety, acceptability and feasibility of delivery of Pre-Exposure Prophylaxis (PrEP) or Post-Exposure Prophylaxis) PEP as part of combination HIV prevention services for high-risk MSM and transgender women.

DETAILED DESCRIPTION:
Two community-based sites (LALGBT Center and The OASIS Clinic) will serve as facilities at which participants may present for screening for prevention services. At the sites, eligibility criteria will be assessed, HIV, Sexually Transmitted Disease (STD) and laboratory testing will be performed, and HIV prevention service referrals will be initiated. Follow-up will be on a monthly basis for the first three months, and then de-escalated to an every-3-month interval.

The program stratifies participants into two cohorts on the basis of sexual risk behavior: a low-moderate risk cohort (LM) and a high-risk cohort (H). Participants in the LM cohort will be provided a customized prevention package (CPP) including access to PEP for emergency HIV prevention in the event of unanticipated HIV exposure. Participants in the H cohort will be provided a CPP including daily Truvada-based PrEP. All participants will be followed for 48 weeks. Participants in the LM cohort who, on longitudinal sexual risk behavior surveillance, report increased levels of sexual risk-taking such that they meet enrollment criteria for the H-cohort will be transitioned to the H-cohort.

At each follow-up visit, a careful safety assessment will be made, including signs/symptoms and laboratory assessments. STD testing will be performed at 3 month intervals. An escalating-intensity adherence intervention will be implemented based on real-time plasma tenofovir levels. A computer-assisted self-interview (CASI) will be used to capture detailed sexual risk, adherence, and substance use behavior.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to understand and provide consent in English or Spanish
* Self identified MSM, MSM/W, or Transfemale
* At least one male sex partner for anal intercourse in the prior 12 months
* HIV negative by enzyme immunoassay (EIA) and viral load (VL)
* CrCl ≥ 60 ml/min (via Cockcroft-Gault formula)
* No signs or symptoms suggestive of primary HIV infection (PHI).

Exclusion Criteria:

* Participants <18 years of age
* Unable to understand and provide consent in English or Spanish
* Known or found on testing to be HIV positive
* Any condition, which in the opinion of the intake provider, will seriously compromise the participant's ability to comply with the protocol, including adherence to PEP or PrEP medication dosing
* Use of Antiretroviral therapy (ART) taken for any indication (i.e. PEP or PrEP) within 60 days of study entry
* Previous participation in an HIV vaccine trial. Participants that were documented to have received only placebo are not excluded.
* Signs or symptoms suspicious for PHI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Landovitz, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - L.A. Gay and Lesbian Center, Los Angeles, California
  - The OASIS Clinic, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 328 participants who enrolled in the study, 27 screen failed for various reasons and were not assigned to a cohort.
Groups:
- Cohort H (PrEP): Participants in the H cohort will be provided with a CPP (customized prevention package) including daily Truvada-based PrEP(Pre-Exposure Prophylaxis).
  High Risk Cohort Criteria (one or more of the following has to be met):
  1. No condom use during anal intercourse with ≥3 male sex partners who are HIV-positive or of unknown HIV status during the last three months.
  2. STI diagnosis during the last 12 months.
  3. Previous PEP use during the last 12 months (* see exclusion criteria)
  4. Has at least one HIV infected sexual partner for ≥4 weeks.
  emtricitabine 200mg/tenofovir 300mg: The intervention medication will be tenofovir + emtricitabine, provided as a fixed-dose combination tablet as Truvada®. Dosing is 1 tablet by mouth once daily. For participants with a a confirmed (i.e. two consecutive) reduction in CrCl to <50 mL/min, Truvada will be dose-reduced to 1 tablet by mouth every other day. For patients with creatinine clearance <30 mL/min, Truvada will be discontinued.
- Cohort LM (PEP): Participants who do not meet criteria for High Risk (Cohort H) will be assigned to the LM (low moderate) cohort and will receive a customized prevention package based on baseline assessments (in the same manner as the Cohort H Participants). In addition, they will receive education on the availability and use of post-exposure prophylaxis.
  emtricitabine 200mg/tenofovir 300mg: The intervention medication will be tenofovir + emtricitabine, provided as a fixed-dose combination tablet as Truvada®. Dosing is 1 tablet by mouth once daily. For participants with a a confirmed (i.e. two consecutive) reduction in CrCl to <50 mL/min, Truvada will be dose-reduced to 1 tablet by mouth every other day. For patients with creatinine clearance <30 mL/min, Truvada will be discontinued.
Period: Overall Study
Arm/Group | Cohort H (PrEP) | Cohort LM (PEP)
Started | 297 | 4
Week 0 | 297 | 4
Week 4 | 284 | 4
Week 8 | 278 | 4
Week 12 | 272 | 2
Week 24 | 260 | 1
Week 36 | 247 | 1
Week 48 | 222 | 1
Completed | 218 | 1
Not Completed | 79 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort H (PrEP) | Cohort LM (PEP) | Total
Number analyzed (Participants) | 297 | 4 | 301
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [28 to 42] | 35 [32 to 39] | 34 [28 to 42]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male: Male | 296 | 4 | 300
  Male: Transfemale | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 150 | 1 | 151
  Non-Hispanic Black | 30 | 0 | 30
  Hispanic/Latino | 82 | 1 | 83
  Asian | 14 | 1 | 15
  Pacific Islander/Alaskan Native | 4 | 0 | 4
  Mixed Race/Other | 16 | 1 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 297 | 4 | 301
Education [Count of Participants; unit: Participants]
  High school or less | 33 | 0 | 33
  Some college | 105 | 1 | 106
  College graduate | 104 | 2 | 106
  Any postgraduate | 55 | 1 | 56
Insurance [Count of Participants; unit: Participants]
  Uninsured | 91 | 2 | 93
  Insured | 200 | 1 | 201
  Unknown | 6 | 1 | 7
Marital Status [Count of Participants; unit: Participants]
  Married/civil union/legal partnership | 9 | 0 | 9
  Living with primary or main partner | 42 | 0 | 42
  Have primary or main partner, not living together | 39 | 0 | 39
  Single/divorced/widowed | 194 | 4 | 198
  Other | 12 | 0 | 12
  Unknown | 1 | 0 | 1
Family Income [Count of Participants; unit: Participants]
  $20,000 or less | 92 | 0 | 92
  $20,001 - $50,000 | 111 | 3 | 114
  $50,001 or more | 94 | 1 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Grade 2 or Higher Adverse Event by Cohort
Description: Number and frequency rate of clinical and laboratory AEs (Gr 2 and above), including SAEs by Cohort.
Time Frame: Baseline to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort H (PrEP) | Cohort LM (PEP)
Number analyzed (Participants) | 297 | 4
Participants | 230 | 0

2. Secondary Outcome: Cohort H PrEP Engagement by Study Visit
Description: Optimal adherence to daily oral emtricitabine/tenofovir disoproxil fumarate by study visit as measured by tenofovir diphosphate (TFV-DP) in dried blood spots (DBS). Optimal adherence is defined as TFV-DP levels great than or equal to 700 femtomoles per punch in DBS samples (approximately 4 or more doses a week over the past 60 days).
Time Frame: Baseline to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort H (PrEP)
Number analyzed (Participants) | 296
Participants
  Week 4 | 246
  Week 12 | 247
  Week 24 | 224
  Week 36 | 212
  Week 48 | 194

3. Other Pre Specified Outcome: Escalation in Transmission Risk Behavior Among Participants Reporting Low Risk Behaviors at Baseline
Description: Changes in sexual risk behavior as assessed via CASI-based self-report questionnaire, measured longitudinally over time.
Time Frame: Baseline to 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Cohort H (PrEP) and Cohort LM (PEP): Participants enrolled in Cohort H (PrEP) and Cohort LM (PEP)
Arm/Group | Cohort H (PrEP) and Cohort LM (PEP)
Number analyzed (Participants) | 301
Participants
  High risk reported at baseline and remained high | 278
  Risk increased from low (baseline) to high | 19
  Low risk reported at baseline and remained low | 4

4. Other Pre Specified Outcome: Number of HIV Seroconversions by Cohort.
Time Frame: Baseline to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort H (PrEP) | Cohort LM (PEP)
Number analyzed (Participants) | 297 | 4
Participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Cohort H (PrEP) | Cohort LM (PEP)
Serious Adverse Events (participants affected / at risk) | 2/297 | 0/4
Other Adverse Events (participants affected / at risk) | 195/297 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort H (PrEP) (N=297) | Cohort LM (PEP) (N=4)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 1 (2) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort H (PrEP) (N=297) | Cohort LM (PEP) (N=4)
Alanine aminotransferase increased (Investigations) | 13 (13) | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 62 (80) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 65 (68) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 84 (109) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 56 (61) | 0 (0)
Syphilis (Infections and infestations) | 33 (35) | 0 (0)
Urethritis chlamydial (Infections and infestations) | 23 (24) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No